CLINICAL TRIAL: NCT01893684
Title: Effects of a Higher Protein Weight Loss Diet and Exercise on Body Composition, Physical Function, and Fatigue in Overweight Older Women
Brief Title: Dietary Intervention and Varying Physical Activity in Seniors
Acronym: ugaDIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Ellen Evans, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCBA; NCBA (Other Grant/Funding Number: National Cattleman's Beef Association)
Record Dates: First submitted 2013-02-04; First posted 2013-07-09 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: protein; physical function; muscle quality; fatigue; weight loss
MeSH Terms: conditions — Obesity; Fatigue; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein + Exercise (Experimental): PRO diet recommendations will include high quality proteins with an emphasis on lean meats, with protein being targeted for every meal and snack. PRO will provide dietary protein (1.6 g.kg-1.d-1; ~30% of energy intake) with a ratio of carbohydrate/protein of <1.5 and dietary lipids at ~ 30% energy intake. Energy deficit will be determined by reducing estimated daily energy needs by ~500 kcal/d. The prescribed diet will include a minimum of one serving of beef per day, which is approximately 3 to 3.5 ounces or ~100 grams. The exercise program will require attendance of 3 nonconsecutive days per week. A program that combines flexibility and balance activities, weight bearing endurance exercise (walking) and resistance training to preserve lean mass will be prescribed. Each session will last ~75 min with a 35 min warm-up/aerobic exercise of mild to moderate intensity, ~30 min of resistance training, and finally, a ~10 min of balance and flexibility exercises during the cool-down period.
  Interventions: Behavioral: Exercise; Behavioral: Higher Protein Diet
- Protein (Experimental): PRO diet recommendations will include high quality proteins with an emphasis on lean meats, with protein being targeted for every meal and snack. PRO will provide dietary protein (1.6 g.kg-1.d-1; ~30% of energy intake) with a ratio of carbohydrate/protein of <1.5 and dietary lipids at ~ 30% energy intake. Energy deficit will be determined by reducing estimated daily energy needs by ~500 kcal/d. The prescribed diet will include a minimum of one serving of beef per day, which is approximately 3 to 3.5 ounces or ~100 grams.
  Interventions: Behavioral: Higher Protein Diet
- Carbohydrate + Exercise (Experimental): Diet will provide dietary protein at 0.8 g.kg-1.d-1 (~ 18% of energy intake) with a ratio of carbohydrates/protein > 3.5 and dietary lipids at ~30% energy intake. Again, energy deficit will be determined by reducing estimated daily energy needs by ~500 kcal/d. The exercise program will require attendance of 3 nonconsecutive days per week. A program that combines flexibility and balance activities, weight bearing endurance exercise (walking) and resistance training to preserve lean mass will be prescribed. Each session will last ~75 min with a 35 min warm-up/aerobic exercise of mild to moderate intensity, ~30 min of resistance training, and finally, a ~10 min of balance and flexibility exercises during the cool-down period.
  Interventions: Behavioral: Exercise; Behavioral: Conventional Carbohydrate Diet

INTERVENTIONS:
Behavioral: Exercise — PRO+EX and CARB+EX groups will be prescribed an exercise program with required attendance of 3 nonconsecutive days per week. Exercise sessions will be supervised and conducted by trained graduate students in the Department of Kinesiology. Based on recommended practice, a program that combines flexibility and balance activities, weight bearing endurance exercise (walking) and resistance training to preserve lean mass will be prescribed. Each session will last ~75 min with a 35 min warm-up/aerobic exercise of mild to moderate intensity, ~30 min of resistance training, and finally, a ~10 min of balance and flexibility exercises during the cool-down period. Endurance training activities will vary but will all be weight-bearing.
  Arms: Carbohydrate + Exercise; Protein + Exercise
Behavioral: Higher Protein Diet — PRO diet recommendations will include high quality proteins with an emphasis on lean meats with protein being targeted for every meal and snack. PRO will provide dietary protein (1.6 g.kg-1.d-1; ~30% of energy intake) with a ratio of carbohydrate/protein of <1.5 and dietary lipids at ~ 30% energy intake. Energy deficit will be determined by reducing estimated daily energy needs by ~500 kcal/d. Regarding beef intake specifically, the prescribed diet will include a minimum of one serving of beef per day, which is approximately 3 to 3.5 ounces or ~100 grams. This amount of lean cooked beef provides an average of ~25-30 grams of protein per day (www.beefnutrition.org/leanbeef.aspx). Our dietary prescription to the PRO groups that they add 3 ounces (and perhaps up to 3.5 ounces pending body size) of lean beef daily will provide an additional 25-30 grams of protein. This diet will also include 5 servings/day of vegetables and 2-3 servings/day of fruit.
  Arms: Protein; Protein + Exercise
Behavioral: Conventional Carbohydrate Diet — For the CARB group, the diet will provide dietary protein at 0.8 g.kg-1.d-1 (~ 18% of energy intake) with a ratio of carbohydrates/protein > 3.5 and dietary lipids at ~ 30% energy intake. Through nutrition education and counseling we will ensure that the CARB group meets the RDA for protein for women of 46 grams per day from a variety of plant and animal sources. Again, energy deficit will be determined by reducing estimated daily energy needs by ~500 kcal/d. Additional recommendations will include 5 servings/day of vegetables and 2-3 servings/day of fruit. Beef intake will be discouraged in the CARB group.
  Arms: Carbohydrate + Exercise

SUMMARY:
The prevalence of obesity continues to increase at an alarming rate for all sectors of the population in the US. Obesity in the older adult cohort is of great concern as it is associated with reductions in mobility, declines in physical performance and increased risk for physical disability. With regard to body composition, a) fat mass has been determined to be a stronger predictor of mobility limitations than low muscle mass in older individuals and alternatively, b) leg lean mass has also been cited as a primary determinant of lower extremity physical function.

Obesity is related to increased levels of fatigue and lack of motivation and mental energy. Fatigue can be categorized as both a subjective perception and a performance decrement. Fatigue can be defined as a perceived lack of physical or mental energy while fatigability is another construct categorized by the degree of fatigue associated with activity in any dimension (i.e. physical, mental, emotional, and/or social).

The impact of a higher protein diet on muscle quality, muscle fatigability, perceptions of fatigue and systemic inflammation in older adults has not been well documented. The utility of a higher protein weight loss diet combined with resistance exercise training to augment fat mass loss, attenuate lean mass loss and improve muscle quality and physical function could potentially be of high value to overweight older women. The potential further benefits of this regimen to enhance mental energy and other aspects of psycho-social well-being are unknown.

The aims of the present study include assessing the effects of the proposed diet and exercise intervention on 1) body composition, 2) strength and muscle quality, and 3) energy and fatigue symptoms.

DETAILED DESCRIPTION:
Our target population includes 75 overweight or obese (BMI >/= 25kg/m^2) women between the ages of 65 and 80.

This study will use a parallel-arm design. After blocking on age and BMI, 75 overweight or obese (BMI ≥ 25 kg/m2) older females (65 - 80 y old) will be randomized into three groups; PRO or CARB diet combined with exercise (PRO+EX;n=25, CARB+EX; n=25) or PRO (n=25) without exercise for 6 months. All groups will have the goal of losing ~10% of initial body weight. We anticipate an adherence rate of 80% (n = 20 in each group remaining). At the initiation of the study, all subjects will be weight stable (within 2 kg) for past 6 mos and sedentary (defined as < 1h/wk or less than 2 exercise sessions per week in the last 6 months). Eligible participants will be planning to live in the community for the duration of the study. Exclusion criteria will include any chronic disease/condition that would not permit exercise or dietary restriction or alter interpretation of data. All subjects will require personal physician clearance prior to enrollment. Main outcome variables of interest are whole body composition, regional body composition, muscle strength endurance and quality, physical function, fatigue and biomarkers related to fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Overweight or obese (BMI ≥ 25 kg/m2)
3. 65-80 years of age
4. English speaking
5. Plan to live in the community for the duration of the study (~6 months)
6. Weight stable (within 2 kg) for the past 6 months
7. Sedentary (defined as <1 hr/week of physical activity or less than 2 exercise sessions per week in the last 6 months)
8. Free of a history or diagnosis of renal insufficiency or disease
9. Willing to obtain physician clearance
10. Willing to be randomized to treatment groups
11. Free of any chronic disease/condition that would not permit exercise or dietary restriction or alter interpretation of data.
12. Willing to meet all study requirements and randomization
13. Non-smoking and tobacco using
14. Able to obtain transportation to the UGA campus

Exclusion Criteria:

1. Normal weight (BMI < 25 kg/m2)
2. Males
3. Dietary restrictions that do not allow for the consumption of beef, as required by our dietary protocol.
4. Weight loss surgery and/or weight loss medications usage.
5. Any metal within the body and claustrophobia which precludes MRI assessment.
6. Mini-mental state exam score < 25
7. Recent or history of unstable CVD
8. Cancer treatment within the last 5 years or active cancer
9. History of lung disease or COPD or severe asthma
10. Use of anti-inflammatory or steroid medications
11. History or severe arthritis or other medical condition that precludes ability to exercise to level needed by study
12. Current diagnosis or history of balance disorders
13. History of mental disorders, dementia, clinical depression or other disorders that preclude adherence to protocols
14. Current weight of 350 pounds of greater, due to weight restrictions on equipment

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Body Composition at 3 Months and 6 Months | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  Abdominal visceral and subcutaneous adiposity and muscle area and adipose infiltration of muscle will be measured using proton-weighted MR imaging. Subjects will be positioned feet first and supine in a 3.0 Tesla whole body imager (Signa, General Electric, Milwaukee, WI, USA). Imaging of the abdominal region and the thigh will be performed with two separate imaging sequences. The following pulse sequence parameters will be used: Fast Spin Echo-XL, TR/TE = 700/8.12 ms; Slice Thickness = 10mm; NEX = 3; Gap thickness = 5mm; ETL = 3; FA = 90; Number of slices = 18; Acquisition Matrix = 320 x 224 (Reconstructed = 512 x 512); FOV = 20cm; Voxel Size = .39 x .39 x 10 mm. Following high resolution T1 imaging, the images will be analyzed to determine the relative amount of fat in images using a modified Dixon method.
  Whole body fat mass, lean mass and bone mass will also be assessed with DXA scanning.
Change from Baseline in Strength & Muscle Quality at 3 Months and 6 Months | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  Using an isokinetic dynamometer (Biodex System Pro 4, Biodex Medical Systems, INC., New York) with the participant positioned according to manufacturer guidelines, four maximal knee extension and knee flexion contractions will be performed and measured at 0, 60 and 180 deg/sec with the testing order (left, right) and velocity (fast, slow, zero) randomized. The isometric (0 deg/sec) effort will be held for 4-seconds. A set of 25 consecutive maximal repetitions at 180 deg/sec will be used to assess muscular endurance.
Change from Baseline in Energy & Fatigue Symptoms/Psychological Function at 3 Months and 6 Months | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  Subjects will take the following battery of psychological questionnaires at three timepoints: Profile of Mood States, Self-Motivation Inventory, Labeled Magnitude Scale, Affect Grid, SF-36, Pittsburgh Sleep Quality Index, Center for Epidemiological Studies Depression Scale, Perceived Stress Scale, WEL Self-Efficacy Questionnaire, Three Factor Eating Questionnaire, Mini-Mental Status, and the Trails B.

SECONDARY OUTCOMES:
Physical Functional Performance | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  A battery of tests will assess multiple components of physical function, including static and dynamic balance, agility, muscular strength and power, and aerobic capacity.
Biomarkers Related to Fatigue | Baseline (Week 0), Post-Intervention (Week 24)
  Fasting blood samples will be obtained and assayed for markers of systemic inflammation [C-reactive protein (CRP) and IL-6] and indicators of anemia (ferritin and vitamin B12) using commercially available ELISA kits samples run in triplicate. Timing for blood sampling for the inflammatory markers will occur greater than 24 but not less than 48 hours post-exercise in the morning after an overnight fast. With the training occurring 3 times per week generally in the morning, this means that if a person exercises on a Monday, their draw will occur on Wednesday prior to that exercise session. This timing also has maximal translational value in that it provides a "snap shot" of our lifestyle intervention. Participants will be queried regarding any acute illnesses during the 48-hours prior to the blood draw and again one week following this laboratory visit to ensure inflammatory status was not falsely elevated.
Physical Activity | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  Physical activity will be quantified using the Physical Activity Scale for the Elderly (PASE) which estimates the total level of household, occupational and leisure-time physical activities. Accelerometers (ActiGraph single-axis model, Health One Technology) will also be used to provide an objective measure of physical activity.
Acceptability | Post-Intervention (Week 24)
  We will use Nominal Group Technique (NGT) as our focus group technique to qualitatively evaluate the interventions. Essentially 2 small groups (10-15 each) within each treatment group will be brought together to generate barriers and facilitations to the program, share ideas and opinions, have a group discussion and then vote and rank major barriers and facilitations to the program. Notably our facilitator will tap both the exercise and diet aspects of our intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Evans, PhD, Principal Investigator — University of Georgia; Rachelle M Acitelli, MS, Study Director — University of Georgia; Chad R Straight, MS, Study Director — University of Georgia; Alison C Berg, MS, RD, Study Director — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

REFERENCES:
- [Derived] Williams ER, Straight CR, Wilson HK, Lynall RC, Gregory CM, Evans EM. Weight Loss and Exercise Effects on Rate of Torque Development and Physical Function in Overweight Older Women. J Aging Phys Act. 2022 Nov 21;31(3):458-464. doi: 10.1123/japa.2022-0032. Print 2023 Jun 1. PMID 36410339
- [Derived] Evans EM, Straight CR, Reed RA, Berg AC, Rowe DA, Johnson MA. Exercise and Protein Effects on Strength and Function with Weight Loss in Older Women. Med Sci Sports Exerc. 2021 Jan;53(1):183-191. doi: 10.1249/MSS.0000000000002429. PMID 32520876
- See also: National Cattleman's Beef Association — http://www.beef.org/
- See also: UGA Department of Kinesiology — http://www.coe.uga.edu/kinesiology/